CLINICAL TRIAL: NCT03641326
Title: Phase II Clinical Trial of Sunitinib in Sarcomas of the Central Nervous System
Brief Title: Sunitinib in Sarcomas of the Central Nervous System
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Gilbert, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180137; 18-C-0137
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Gliosarcoma; Central Nervous System Sarcoma
Keywords: Gliosarcoma; Brain Tumor; MDASI
MeSH Terms: conditions — Gliosarcoma; Brain Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Participants With Primary Gliosarcoma (Experimental): Sunitinib will be administered at a dose of 50 mg daily for 2 consecutive weeks followed by 1 week of rest. Participants will be given a small, portable pager-type and watch accelerometers to wear at the hip or non-dominant wrist. Worn daily for 6 cycles
  Interventions: Drug: Sunitinib; Device: wGT3x-BT
- Participants With Secondary Gliosarcoma (Experimental): Sunitinib will be administered at a dose of 50 mg daily for 2 consecutive weeks followed by 1 week of rest. Participants will be given a small, portable pager-type and watch accelerometers to wear at the hip or non-dominant wrist. Worn daily for 6 cycles
  Interventions: Drug: Sunitinib; Device: wGT3x-BT
- Participants With Primary Central Nervous System (CNS) Sarcoma (Experimental): Sunitinib will be administered at a dose of 50 mg daily for 2 consecutive weeks followed by 1 week of rest. Participants will be given a small, portable pager-type and watch accelerometers to wear at the hip or non-dominant wrist. Worn daily for 6 cycles
  Interventions: Drug: Sunitinib; Device: wGT3x-BT

INTERVENTIONS:
Drug: Sunitinib — Sunitinib will be administered at a dose of 50 mg daily for 2 consecutive weeks followed by 1 week of rest until there is disease progression or development of intolerable side effects.
  Other Names: Sutent
Device: wGT3x-BT — Participants will given a small, portable pager-type and watch accelerometers to wear at the hip or non-dominant wrist. Worn daily for 6 cycles
  Other Names: Actigraph

SUMMARY:
Background:

A sarcoma is a rare cancer. It grows in the body's connective tissue. Sarcomas in the brain and central nervous system are especially rare. The drug Sunitinib has been approved in many countries for treating other types of rare or advanced cancers. These include kidney, pancreas, and bowel cancer. Researchers want to see if it can help people with sarcomas of the central nervous system.

Objective:

To study the effects of Sunitinib on gliosarcomas or sarcomas of the central nervous system.

Eligibility:

Adults ages 18 and older with a gliosarcoma or sarcoma of the central nervous system

Design:

Participants will be screened with the following tests. Some may be done as part of their regular cancer care:

Medical history

Medication review

Physical exam

Blood, heart, and pregnancy tests

Cranial scans to locate and measure their tumor

Participants will take Sunitinib by mouth every day for 2 weeks and then take none of the drug for 1 week. These 3 weeks equal 1 cycle.

Participants will have 2 study visits in cycle 1. They will have 1 visit in all other cycles. They will answer questions about quality of life and repeat some screening tests.

Participants will take their blood pressure at home weekly. They keep a diary of each dose of Sunitinib and blood pressure reading.

Participants can choose to share data about their physical activity levels and quality of sleep. These participants will wear a small, portable watch-sized accelerometer device on the wrist for 6 cycles.

About 1 month after their last study drug dose, participants will have a final study visit. They will have a physical exam, blood tests, and scans.

DETAILED DESCRIPTION:
Background:

* Gliosarcoma and primary central nervous system (CNS) sarcomas are malignant brain tumors uniformly associated with poor outcome.
* There are no known effective medical therapies for these cancers.
* Sunitinib is an orally administered small molecule that inhibits signaling of multiple receptor tyrosine kinases including those known to be activated in CNS sarcomas.

Objectives:

To determine the anti-tumor effect of sunitinib in recurrent gliosarcomas and primary CNS sarcomas as assessed by objective response rate (ORR).

Eligibility:

* Patients with histologically proven gliosarcoma and primary CNS sarcoma at disease relapse after failing standard therapy (surgery and irradiation).
* Tumor tissue blocks or 15 unstained slides should be available
* Subjects must be greater than or equal to 18 years old.
* Karnofsky performance status of greater than or equal to 60
* Patients must have adequate organ function.
* Patients must not have received tyrosine kinase inhibitor(s) in the past.

Design:

* This is a prospective, single institution, single arm, multi-cohort phase II study of sunitinib in subjects with recurrent gliosarcoma and primary CNS sarcoma that have failed prior surgery and irradiation (unless radiation therapy was contraindicated).
* Subjects will be classified into three cohorts: 1) Primary gliosarcoma; 2) Secondary gliosarcoma; 3) Primary CNS sarcoma. Cohort expansion will be carried out at indication of promising response.
* Sunitinib will be administered orally using a continuous schedule at 50 mg per day (with dose adjustments allowed for toxicity) for 2 weeks with 1 week off to constitute a 3-week cycle until disease progression or development of intolerable side-effects.
* Toxicity will be assessed every cycle by Common Terminology Criteria in Solid Tumors (CTCAE) version 5.0.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed gliosarcoma (primary or secondary) or primary central nervous system sarcoma confirmed by the Laboratory of Pathology, National Cancer Institute (NCI).
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured bi-dimensionally by MRI (or computed tomography (CT) scan if magnetic resonance imaging (MRI) is contraindicated).
* Patients must have failed standard therapy consisting of surgery, irradiation, and chemotherapy if indicated.
* Age greater than or equal to 18 years.
* Karnofsky greater than or equal to 60%.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with

creatinine levels above institutional normal.

* Patients must have the ability to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of this study.
* The effects of sunitinib on the developing human fetus are unknown. For this reason and because anti-angiogenic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Tumor tissue blocks or at least 10-15 unstained slides from the diagnosis should be available.
* At the time of registration, all subjects must be removed greater than or equal to 28 days from any investigational agents.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior use of tyrosine kinase inhibitors or vascular endothelial growth factor (VEGF) inhibition.
* Patients who are receiving strong cytochromes P450 (CYP450) inducers or inhibitors are ineligible.
* Pregnant women are excluded from this study because sunitinib has potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib, breastfeeding should be discontinued if the mother is treated with sunitinib.
* Patients with known human immunodeficiency virus (HIV) history on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with sunitinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Uncontrolled hypertension (> 150/100 mm hemoglobin (Hg) while on antihypertensive medications.
* New York Heart Association class II or greater congestive heart failure.
* Serious cardiac arrhythmia requiring medication.
* Baseline echocardiogram with ejection fraction < 50% or greater than or equal to 20% decrease from a prior study.
* Corrected QT interval (QTc) > 500 msec on baseline electrocardiogram (EKG)
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis. Note: Low molecular weight heparin is permitted provided the patient's international normalized ratio (INR) is less than or equal to 1.5.
* Previous exposure to anthracyclines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Gilbert, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kondo T, Takagi T, Kobayashi H, Iizuka J, Nozaki T, Hashimoto Y, Ikezawa E, Yoshida K, Omae K, Tanabe K. Superior tolerability of altered dosing schedule of sunitinib with 2-weeks-on and 1-week-off in patients with metastatic renal cell carcinoma--comparison to standard dosing schedule of 4-weeks-on and 2-weeks-off. Jpn J Clin Oncol. 2014 Mar;44(3):270-7. doi: 10.1093/jjco/hyt232. Epub 2014 Jan 27. PMID 24474815
- [Background] Cachia D, Kamiya-Matsuoka C, Mandel JJ, Olar A, Cykowski MD, Armstrong TS, Fuller GN, Gilbert MR, De Groot JF. Primary and secondary gliosarcomas: clinical, molecular and survival characteristics. J Neurooncol. 2015 Nov;125(2):401-10. doi: 10.1007/s11060-015-1930-y. Epub 2015 Sep 9. PMID 26354773
- [Background] Finke J, Ko J, Rini B, Rayman P, Ireland J, Cohen P. MDSC as a mechanism of tumor escape from sunitinib mediated anti-angiogenic therapy. Int Immunopharmacol. 2011 Jul;11(7):856-61. doi: 10.1016/j.intimp.2011.01.030. Epub 2011 Feb 11. PMID 21315783
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0137.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants with Primary Central Nervous System (CNS) Sarcoma were enrolled in Cohort 3.
Groups:
- Participants With Primary Gliosarcoma; Participants With Secondary Gliosarcoma: Sunitinib administered orally using a continuous schedule at 50 mg per day (with dose adjustments allowed for toxicity) for 2 weeks with 1 week off to constitute a 3-week cycle until disease progression or development of intolerable side-effects.
Period: Overall Study
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (12.45) | 58.6 (10.16) | 62.24 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Greater Than 50% Reduction in Objective Response
Description: Objective Response is defined as all participants who had greater than 50% reduction in Complete Response and Partial Response assessed by the Assessment in Neuro-oncology Criteria (RANO criteria). Complete Response is no T1 gadolinium enhancing disease, no new lesions, or corticosteroids, and stable or decreasing T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) or clinical status. Partial Response is ≥50% decrease in T1 gadolinium enhancing disease, no new lesions, stable or decreasing T2/FLAIR or corticosteroids, and stable or increasing clinical status.
Time Frame: From enrollment to off study, approximately 3 Months, 1 Week, 4 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
Number analyzed (Participants) | 2 | 3
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

2. Secondary Outcome: Number of Participants With 6-month Progression Free Survival (PFS)
Description: Progression is defined as the duration of time from start of treatment to time of progression or death, whichever comes first. PFS was assessed by the Response Assessment in Neuro-oncology Criteria (RANO criteria). Progression is ≥25% increase in T1 gadolinium enhancing disease, increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR), presence of new lesions, and decrease in clinical status.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

3. Secondary Outcome: Number of Participants That Have Progressive Disease After 18 Months
Description: Progressive disease was assessed by the Response Assessment in Neuro-oncology Criteria (RANO criteria). Progression is ≥25% increase in T1 gadolinium enhancing disease, increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR), presence of new lesions, and decrease in clinical status.
Time Frame: After 18 months
Population: This outcome measure was not analyzed because none of the participants reached 6 months progression free survival (PFS), thus we could not assess participants for 18 months PFS.
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Adverse Events Related to Drug
Description: Adverse events was assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Baseline to off study, approximately 3 months and 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

5. Secondary Outcome: Evaluation of Tumor Tissue for Biomarkers
Description: To evaluate archival tumor tissue for activation of signaling pathways targeted by sunitinib to establish potential biomarkers of response.
Time Frame: end of study, approximately 25 months and 12 days.
Population: Analysis not done. There were not enough samples collected to provide results.
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Responders and Non-responders With Tumor Markers of Activation
Description: Molecular profiling of archival tumor tissues was used to identify tumor markers of activation of response to sunitinib in responders and non-responders. A responder is a participant with a Complete Response (CR) or Partial Response (PR), and a non-responder is a participant with Stable Disease (SD) or Progressive Disease (PD) assessed by the Response Assessment in Neuro-oncology Criteria (RANO criteria). CR is no T1 gadolinium enhancing disease, no new lesions, or corticosteroids, and stable or decreasing T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR). PR is ≥50% decrease in T1 gadolinium enhancing disease, no new lesions, stable or decreasing T2/FLAIR or corticosteroids, and stable or increasing clinical status. SD is <50% decrease in T1 gadolinium enhancing disease but < 25% increase, no new lesions, stable or decreasing T2/FLAIR or corticosteroids, and stable or increase in clinical status. PD is ≥25% increase in T1 gadolinium enhancing disease.
Time Frame: From baseline to end of treatment, approximately 25 months and 12 days.
Population: 0 participants achieved a response in the responders with primary gliosarcoma group and responders with secondary gliosarcoma group.
Measure: Count of Participants; unit: Participants
Groups:
- Responders With Primary Gliosarcoma; Responders With Secondary Gliosarcoma: A responder is a participant with a Complete Response (CR) or Partial Response (PR).
- Non-Responders With Primary Gliosarcoma; Non-Responders With Secondary Gliosarcoma: A non-responder is a participant with Stable Disease (SD) or Progressive Disease (PD).
Arm/Group | Responders With Primary Gliosarcoma | Non-Responders With Primary Gliosarcoma | Responders With Secondary Gliosarcoma | Non-Responders With Secondary Gliosarcoma
Number analyzed (Participants) | 0 | 2 | 0 | 3
Participants | 0 | 1 | 0 | 2

7. Secondary Outcome: Number of Responders and Non-responders With a Change in Perfusion Blood Volume Before and After Treatment With Sunitinib.
Description: Perfusion was quantitated in responders and non-responders comparing pre and post treatment to determine if the treatment regimen altered vasculature and blood flow to the tumor. A responder is a participant with a Complete Response (CR) or Partial Response (PR), and a non-responder is a participant with Stable Disease (SD) or Progressive Disease (PD) assessed by the Response Assessment in Neuro-oncology Criteria (RANO criteria). CR is no T1 gadolinium enhancing disease, no new lesions, or corticosteroids, and stable or decreasing T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR). PR is ≥50% decrease in T1 gadolinium enhancing disease, no new lesions, stable or decreasing T2/FLAIR or corticosteroids, and stable or increasing clinical status. SD is <50% decrease in T1 gadolinium enhancing disease but <25% increase, no new lesions, stable or decreasing T2/FLAIR or corticosteroids, and stable or increase in clinical status. PD is ≥25% increase in T1 gadolinium enhancing disease.
Time Frame: Pre-treatment and post treatment, approximately 25 months and 12 days.
Population: This outcome measure was not done because no data was collected because the perfusion blood volume was not measured.
Arm/Group | Responders With Primary Gliosarcoma | Non-Responders With Primary Gliosarcoma | Responders With Secondary Gliosarcoma | Non-Responders With Secondary Gliosarcoma
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Responders and Non-responders With Dynamic Contrast Enhanced Magnetic Resonance Imaging (MRI) Performed Before and During Treatment With Sunitinib.
Description: Dynamic contrast enhanced magnetic resonance imaging (MRI) was performed before and during treatment with sunitinib in responders and non-responders. A responder is a participant with a Complete Response (CR) or Partial Response (PR), and a non-responder is a participant with Stable Disease (SD) or Progressive Disease (PD) assessed by the Response Assessment in Neuro-oncology Criteria (RANO criteria). CR is no T1 gadolinium enhancing disease, no new lesions, or corticosteroids, and stable or decreasing T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR). PR is ≥50% decrease in T1 gadolinium enhancing disease, no new lesions, stable or decreasing T2/FLAIR or corticosteroids, and stable or increasing clinical status. SD is <50% decrease in T1 gadolinium enhancing disease but < 25% increase, no new lesions, stable or decreasing T2/FLAIR or corticosteroids, and stable or increase in clinical status. PD is ≥25% increase in T1 gadolinium enhancing disease.
Time Frame: Before (baseline) and during treatment with Sunitinib every 6 weeks, up to approximately 25 months and 12 days.
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Responders With Primary Gliosarcoma | Non-Responders With Primary Gliosarcoma | Responders With Secondary Gliosarcoma | Non-Responders With Secondary Gliosarcoma
Number analyzed (Participants) | 0 | 2 | 0 | 3
Participants
  Baseline | 0 | 2 | 0 | 3
  During Treatment: number analyzed (Participants) | 0 | 1 | 0 | 2
  During Treatment | 0 | 1 | 0 | 2

9. Secondary Outcome: Mean Symptom Severity and Interference From Baseline Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT)
Description: Participants reported outcome measures using a self-reported symptom severity and interference with daily activities using the MDASI-BT. The MDASI-BT consists of symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. All patients with at least one valid questionnaire will be included in the analyses. This outcome measure was predicated on change. Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom severity and symptom interference measures.
Time Frame: Baseline and off treatment, approximately 25 months and 12 days
Population: 2 participants only had baseline MDASI, & 1 participant had baseline&off treatment MDASI in the secondary glioblastoma group. The number of participants enrolled =5 & analyses were performed on a subset of collected data. No conclusions should be drawn from the reported data on whether participants had a change in quality of life. Only treatment toxicity evaluation is meaningful & this will not vary by the histologic subtype of the tumor. Thus, combining the 2 groups is most logical & expedient.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Participants With Primary Gliosarcoma and Secondary Gliosarcoma: Sunitinib administered orally using a continuous schedule at 50 mg per day (with dose adjustments allowed for toxicity) for 2 weeks with 1 week off to constitute a 3-week cycle until disease progression or development of intolerable side-effects.
Arm/Group | Participants With Primary Gliosarcoma and Secondary Gliosarcoma
Number analyzed (Participants) | 2
Score on a scale
  Baseline mean symptom severity | 2.4 (1.5)
  Baseline mean symptom interference | 3.4 (3.4)
  Mean symptom severity at disease progression: number analyzed (Participants) | 1
  Mean symptom severity at disease progression | 0.4 (NA) — Standard Deviation cannot be calculated at disease progression due to n=1.
  Mean symptom interference at disease progression: number analyzed (Participants) | 1
  Mean symptom interference at disease progression | 0.2 (NA) — Standard Deviation cannot be calculated at disease progression due to n=1.

10. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Baseline to off study, approximately 3 months and 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Baseline to off study, approximately 3 months and 12 days
Arm/Group | Participants With Primary Gliosarcoma | Participants With Secondary Gliosarcoma
All-Cause Mortality (participants affected / at risk) | 2/2 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/2 | 3/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Primary Gliosarcoma (N=2) | Participants With Secondary Gliosarcoma (N=3)
Edema face (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Nervous system disorders - Other, Apraxia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Primary Gliosarcoma (N=2) | Participants With Secondary Gliosarcoma (N=3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (2)
General disorders and administration site conditions - Other, bilateral feet ache (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (4)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (8) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (6)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, apraxia (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Yellowing skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
National Institutes of Health (NIH) clinical center is a quaternary care facility where we rely heavily on self-referrals and outside physician referrals for accrual. Competing trials at NIH and outside institutions have shifted interest from this study and physicians are not referring patients for this study. Consequently, we have had low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03641326/Prot_SAP_002.pdf
  • Informed Consent Form (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03641326/ICF_001.pdf